CLINICAL TRIAL: NCT01589029
Title: A Pilot Study on the Effects of ILARIS® on Patients With Proliferative Diabetic Retinopathy (PDRP)
Acronym: ILARIS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The results of the interim analysis showed that the primary endpoint was not met
Sponsor: PD Dr. med. Stephan Michels (Other)
Collaborators: Novartis (Industry); University Hospital, Zürich (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Stephan Michels, Stephan Michels, MD, MBA, Associate Professor, Head Medical Retina, Department of Ophthalmology, Triemli Hospital, Triemli Hospital
Organization: Triemli Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885MCH01T
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CANAKINUMAB (ILARIS®) (Other)
  Interventions: Drug: CANAKINUMAB (ILARIS®)

INTERVENTIONS:
Drug: CANAKINUMAB (ILARIS®) — subcutaneous injection every 8 weeks

SUMMARY:
The pilot study evaluates the efficacy and safety of Canakinumab (ILARIS®) in subjects with proliferative diabetic retinopathy secondary to type 1 and 2 diabetes. Ten subjects will be enrolled to receive 150 mg Canakinumab (ILARIS®) by subcutaneous injection. Beginning on day 0, each subject will receive a subcutaneous injection of study drug every 8 weeks for 16 weeks, a total of 3 injections. All subjects will undergo regular follow-up assessments every 8 weeks through 24 weeks. Fluorescein angiography (FA) is repeated every 8 weeks. In case of progression of retinal neovascularization on FA panretinal laser photocoagulation is administered as rescue therapy. The primary outcome is the regression of retinal neovascularizations (NVE and NVD) in FA at 24 weeks. In addition to key secondary outcomes including regression of diabetic macular edema, change in best-corrected visual acuity, change in HbA1c levels and change in markers of systemic inflammation. Safety will be assessed by measurements of vital signs, clinical laboratory assessments, and the recording of adverse clinical events.

ELIGIBILITY:
Inclusion Criteria:

Signed and dated Informed Consent

American Diabetes Association (ADA) diagnostic criteria for type 1 (TD1) or type 2 (T2D) diabetes

Evidence of proliferative diabetic retinopathy with:

1. Active retinal neovascularization defined by fluorescein angiography as non-high risk proliferative diabetic retinopathy (PDRP; NVD < 1/3 disc area; NVE < ½ disc area) or
2. High risk PDRP treated with prior panretinal laser photocoagulation (PRP), showing persistent, active retinal neovascularization. The last session of PRP should not be within 12 weeks prior to enrolment.

Diabetes (Type I or II) must be stable which is defined as not requiring a change in medication over the last 4 weeks

Age ≥ 18

For female subjects of child-bearing age, a negative serum pregnancy test is mandatory. For subjects with reproductive potential, a willingness to utilize adequate contraception and not become pregnant. Adequate contraceptive measures include oral contraceptives (stable use for two or more cycles prior to Screening); IUD; Depo-Provera®; Norplant® System implants; condom or diaphragm used in conjunction with contraceptive sponge, foam or jelly; and abstinence.

Ability to regular follow-up visits

-

Exclusion Criteria:

Patients requiring laser coagulation or intravitreal therapy with steroids or anti-VEGF drugs for diabetic macular edema within the first 6 months after enrolment

Patients with laser coagulation or any intravitreal therapy within three months prior to enrollment Media opacification not allowing adequate retinal examination

Allergy to fluorescein (Fluorescein Angiography)

Known HIV antibody, hepatitis B surface antigen, and/or hepatitis C antibody

History of malignancy except basal cell skin carcinoma prior to study entry

History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody

History or evidence of active tuberculosis (TB) infection at Visit 1 or one of the risk factors for tuberculosis such as residence in a congregate setting (e.g. homeless shelter), substance abuse, health-care workers with unprotected exposure to patients who are at high risk of TB or patients with TB disease, close contact (i.e. share the same air space in a household or other enclosed environment for a prolonged period (days or weeks) with a person with active pulmonary TB disease within the last 12 months

History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection, at Visit 1, determined as defined by local guidelines/ local medical practice. If presence of tuberculosis is established then treatment (according to local guidelines) must have been completed prior to randomization

Live vaccinations within 3 months prior to the randomization visit or live vaccinations planned during the trial.

History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes

Any biologic drugs targeting the immune system (for example, TNF blockers, anakinra, rituximab, abatacept, tocilizumab)

active atopic disease

history or symptoms of a demyelinating disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Regression of retinal neovascularizations (NVE and NVD) in FA. | 24 weeks

SECONDARY OUTCOMES:
Central retinal thickness measured by SD-OCT | 24 weeks
Best corrected visual acuity | 24 weeks
Change in HbA1c and inflammatory markers | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Michels, MD, MBA, Principal Investigator — Department of Ophthalmology, Triemli Hospital Zuerich
Locations (1):
- Department of Ophthalmology, Triemli Hospital Zurich, Zurich, Canton of Zurich, Switzerland